CLINICAL TRIAL: NCT05398068
Title: Effects of Exercise Training on Exercise Capacity and Sleep Quality in Patients With Obesity Hypoventilation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proffesor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/30
Record Dates: First submitted 2022-05-22; First posted 2022-05-31 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity Hypoventilation Syndrome (OHS); Hypoventilation; Obesity; Respiration Disorders; Sleep Disorder
Keywords: Obesity; Exercise Capacity; Physical Activity; Quality of Life; Hand Grip Strength; Anxiety; Depression
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Hypoventilation; Obesity; Respiration Disorders; Sleep Wake Disorders; Motor Activity; Anxiety Disorders; Depression | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training (Exercises and Diet) Group (Experimental): Training (Exercises and Diet) Group; Patients will follow a regular diet program for 10 weeks.
  Aerobic exercises will be planned for patients 2 days a week under the supervision of a physiotherapist, and 3 days a week as home exercises.
  Strengthening exercises will be planned for patients 1 days a week under the supervision of a physiotherapist, and 2 days a week as home exercises.
  Interventions: Other: Exercises and Diet
- Control (Diet) Group (Active Comparator): Control (Diet) Group; Patients will follow a regular diet program for 10 weeks.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Exercises and Diet — Non-Invasive Ventilation (NIV) will be included in the treatment program of all patients participating in the study. For the Mediterranean diet protocol planned in training groups; each patient will be evaluated by a dietitian at the beginning of the study and individual diet programs will be planned.
  A 10-week exercise training will be planned for the training group.
  Aerobic exercise sessions will be planned as a 5-minute warm-up - 20-minute bicycle ergometer - 5-minute cooling-down program. The intensity of exercise will be planned to be of medium intensity according to the heart rate reserve (40-50%). According to the Modified Borg Scale, walking will be given 3 days a week at a intensity of 4-6, also as a home exercise.
  Strengthening exercises will be planned with reference to 10 RM (repetition maximum) with theraband for large muscle groups (10 repetitions-3 sets).
  Arms: Training (Exercises and Diet) Group
Other: Diet — Non-Invasive Ventilation (NIV) will be included in the treatment program of all patients participating in the study. A regular diet program will be planned for 10 weeks for the control group. . For the Mediterranean diet protocol planned in control groups; each patient will be evaluated by a dietitian at the beginning of the study and individual diet programs will be planned. After that, after 1 week, patients will be re-evaluated for compliance by a dietitian. And than, each patient included in the study will be evaluated for 2 weeks during the treatment period.
  Arms: Control (Diet) Group

SUMMARY:
Obesity Hypoventilation Syndrome is defined as a combination of obesity (BMI ≥ 30 kg/m2) and daytime hypercapnia in arterial blood gas analysis (PaCO2 > 45 mmHg) without other pathologies that cause hypoventilation. Symptoms seen in individuals diagnosed with OHS are stated as a feeling of suffocation due to apnea, loud snoring, morning headache and excessive daytime sleepiness. Respiratory mechanics, respiratory muscle performance, pulmonary gas exchange, lung functions and exercise capacity parameters are adversely affected in patients. Early treatment is important so that these negative changes do not lead to worse outcomes. Weight control, bariatric surgery, pharmacological treatment and non-invasive mechanical ventilation (NIMV) are included in the treatment program of OHS patients. The effects of exercise on the treatment program of OHS patients are unknown. Considering all the studies in the literature, the primary purpose of this study is to evaluate aerobic and strength training on exercise capacity and sleep quality in patients with hypoventilation syndrome. The secondary aim is to examine the effect of this exercise training on peripheral muscle strength, emotional state, body composition and quality of life parameters. In addition, the researchers believe that this study will form the basis for further scientific studies on OHS and exercise and will make an important contribution to the literature.

DETAILED DESCRIPTION:
Patients with Obesity Hypoventilation Syndrome followed for at least 1 month in the Department of Chest Diseases, Faculty of Medicine, Istanbul University will be included in the study. The patients will be divided into two groups using the computer-assisted randomization program as the study and control groups. The study will be conducted in accordance with the Declaration of Helsinki and consent form will be obtained from the patients participating in the study, indicating that they are willing to participate in the study. Before starting the study, the purpose of the study will be explained to the participants and all information about the study will be given. After 10 weeks of exercise training, patients will be evaluated with, Six-Minute Walking Test, pittsburgh sleep quality index, Body Composition, Nottingham Health Profile, Hospital Anxiety and Depression Scale and Muscle strength. The primary aim is to examine the effects of evaluate aerobic and strengthening training on exercise capacity and sleep quality in patients with hypoventilation syndrome. The secondary aim is to examine the effect of this exercise training on peripheral muscle strength, emotional state, body composition and quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients who have been diagnosed with Obesity Hypoventilation Syndrome

Exclusion Criteria:

* Patients who participate in any other diet program
* Patients who are incompatible with a diet program or exercise program
* Patients with uncontrollable respiratory and comorbid diseases
* Patient who have been an orthopedic, neurological, cardiac, or metabolic condition that may prevent participation and continuation of the exercise program throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Six Minutes Walk Test | 10 weeks
  The distance covered in meters in a straight corridor of 30 meters will be recorded as fast as possible but without running for 6 minutes. The distance that normal individuals should take in this period is 400-700 meters. In addition, oxygen saturation and heart rate, resting fatigue and dyspnea levels will be evaluated with pulse oximetry before and after testing. Modified Borg Dyspnea and Fatigue Scales will be used to determine resting dyspnea and fatigue levels.
Pittsburgh Sleep Quality Index | 10 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders. Clinical studies have found the PSQI to be reliable and valid in the assessment of sleep problems to some degree, but more so with self-reported sleep problems and depression-related symptoms than actigraphic measures.
Epworth Sleepiness Scale | 10 weeks
  The Epworth Sleepiness Scale is designed to assess the tendency to fall asleep during the day and the frequency of such episodes. It consists of eight different situations in which participants rate their likelihood of dozing off. Each item is scored on a 4-point scale ranging from 0 to 3, resulting in a total score between 0 and 24. A total score greater than 10 indicates excessive daytime sleepiness.

SECONDARY OUTCOMES:
Nottingham Health Profile | 10 weeks
  The Nottingham Health Profile (NHP) is a general patient reported outcome measure which seeks to measure subjective health status. It is a questionnaire designed to measure a patient's view of their own health status, in a number of areas. The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. The second part of the NHP is optional and can be omitted without ruining the test results.
Hospital Anxiety and Depression Scale | 10 weeks
  7 items of the scale assess anxiety and 7 items assess depression. The answers, which are evaluated in a three-point Likert format, are scored between 0-3. When patients scored 0-10 for anxiety, patients were defined as no anxiety, 11 or more anxiety, and 0-7 points for depression as no depression, 8 or more depression.
Muscle Strength - Dynamometer | 10 weeks
  A digital dynamometer will be used to evaluate muscle strength. Muscle strength will be evaluated in the following muscles, each measurement will be made three times and the average will be taken.
Body Fat Percentage | 10 weeks
  The body fat percentage of a patient is the total mass of fat divided by total body mass, multiplied by 100; body fat includes essential body fat and storage body fat. The body fat percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in percent.
Body Fluid Percentage | 10 weeks
  Body fluids, bodily fluids, or biofluids are liquids within the human body. The body fluid percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in percent.
Muscle Mass | 10 weeks
  Muscle mass refers to the amount of soft muscle tissue in the body. The muscle mass of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results will be recorded in kg.
Body Mass Index | 10 weeks
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Handgrip Strength | 10 weeks
  Handgrip strength will be assessed using a Jamar Hydraulic Hand Dynamometer (USA). The dominant hand will be used as reference. Before each evaluation, the dynamometer will be calibrated. Participants will be seated in an upright position with the arm adducted, elbow flexed at 90°, forearm in neutral position, and the wrist positioned at approximately 30° extension and 5° ulnar deviation, supported on a surface. During each trial, participants will be instructed to squeeze the dynamometer with maximum effort for 5 seconds. Three consecutive measurements will be obtained, with 30-second rest intervals to minimize fatigue. The mean value of the three trials will be recorded in pounds (lb).
Physical Activity Level | 10 weeks
  Physical activity level will be assessed using a pedometer (Hattrick PD-30, China). The device is a portable, cost-effective, and easily accessible motion-sensor tool that records various physical activity parameters, including step count, walking speed, calories expended, and distance walked. In this study, the pedometer will be used to record daily step count, calories burned, and walking distance. The device has the capacity for daily recordings only.
Neck Circumference | 10 weeks
  Neck circumference will be measured with a non-elastic tape measure, recorded in centimeters (cm). Measurements will be performed while the participant is standing upright with weight evenly distributed on both feet. The measurement point will be taken just below the larynx.
Waist circumference | 10 weeks
  Waist circumference will be measured with a non-elastic tape measure, recorded in centimeters (cm). Measurements will be performed while the participant is standing upright with weight evenly distributed on both feet. The measurement point will be the midpoint between the lower margin of the last rib and the top of the iliac crest.
Hip circumference | 10 weeks
  Hip circumference will be measured with a non-elastic tape measure, recorded in centimeters (cm). Measurements will be performed while the participant is standing upright with weight evenly distributed on both feet. The measurement point will be taken at the level of the greater trochanter of the femur.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No